CLINICAL TRIAL: NCT02190591
Title: Use of Peanut Labor Ball for Pelvic Positioning for Nulliparous Patients Following Epidural
Brief Title: Use of Peanut Labor Ball Following Epidural Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Principal Investigator, Rachel Baker, Nurse Researcher, TriHealth Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 14034-14-027
Record Dates: First submitted 2014-05-16; First posted 2014-07-15 (Estimated); Results first posted 2016-11-25 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-03

CONDITIONS: Pregnancy
Keywords: epidural; pregnant; Cesarean Section; forceps; vaginal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pillow and Wedge (No Intervention): Receiving standard care for positioning during labor using pillows and wedges
- Peanut Labor Ball (Experimental): Use of the peanut labor ball within 30 minutes after epidural placement
  Interventions: Device: Peanut Labor Ball

INTERVENTIONS:
Device: Peanut Labor Ball — Peanut Labor Ball
  Arms: Peanut Labor Ball

SUMMARY:
The purpose of the study is to look at the impact of using the Peanut Labor Ball (PLB) after epidural anesthesia in patients who have never given birth. The study will measure the impact on the length of labor, cesarean section rate, operative vaginal delivery rate (vacuum or forceps use), and third or fourth degree laceration rates. This study will determine the impact of PLB use by comparing two cohorts of nulliparous patients: one with the PLB use and one with traditional wedge and pillow positioning. If benefits related to use of the PLB can be demonstrated, it is our intention that each labor room will be stocked with a PBL for use as standard of care.

This study will test the following hypotheses:

1. The Peanut Labor Ball (PLB) will impact the cesarean section and operative vaginal delivery rate in low risk nulliparous patients who receive epidural anesthesia compared to similar cohort using traditional wedge and pillow positioning.
2. Using the PLB will impact the amount of time from epidural placement to complete dilation and the time of second stage of labor, when compared with the control cohort.
3. Use of the PLB will impact the third and fourth degree laceration rates when compared with the control cohort.

DETAILED DESCRIPTION:
See above

ELIGIBILITY:
Inclusion Criteria:

* Any nulliparous woman age ≥18 years presenting in labor (or for induction of labor) with:

Gestation: 37 0/7weeks- 41 6/7weeks -early, full, and late term gestations (ACOG, 2013).

* Single gestation
* Vertex presentation
* Plans to deliver with epidural anesthesia

Exclusion Criteria:

* A complication of pregnancy at the time of admission (including known fetal anomalies or placental anomalies)
* Any muscular or skeletal limitations of the patient that does not allow for positioning with the peanut labor ball (PLB)
* An inability to speak or understand English language
* Preterm gestation: <36 6/7 weeks or Post-term >42 0/7weeks
* A multiple gestation
* Non-vertex presentation
* Diabetes including Gestational Diabetes Mellitus (GDM)
* Order for magnesium sulfate infusion
* Plan for delivery without epidural
* Planned cesarean delivery

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 204 (Actual)
Dates: Start 2014-05; Primary Completion 2014-12 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Evans, RN, Principal Investigator — TriHealth Inc.
Locations (1):
- Good Samaritan TriHealth Hosptial, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 204 patients were enrolled between 5/22/2014 and 12/23/2014
Period: Overall Study
Arm/Group | Pillow and Wedge | Peanut Labor Ball
Started | 102 | 102
Completed | 100 | 91
Not Completed | 2 | 11
Not completed — Withdrawal by Subject | 1 | 8
Not completed — Protocol Violation | 1 | 0
Not completed — did not use peanut ball as instructed | 0 | 2
Not completed — face presentation so she was ineligible | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pillow and Wedge | Peanut Labor Ball | Total
Number analyzed (Participants) | 100 | 91 | 191
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.5 (4.7) | 26.7 (4.9) | 26.6 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 91 | 191
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 100 | 91 | 191

OUTCOME MEASURES:

1. Primary Outcome: Delivery Rate
Description: Rate of patients who deliver by cesarean section
Time Frame: .5-72 hours
Measure: Number; unit: participants
Arm/Group | Pillow and Wedge | Peanut Labor Ball
Number analyzed (Participants) | 100 | 91
participants | 31 | 21

2. Secondary Outcome: Dilation to Second Stage Labor
Description: Examining if use of the peanut labor ball has an effect on time between administration of epidural to complete dilation
Time Frame: thirty minutes after epidural given to birth of baby
Population: Included participants with vaginal delivery only
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Pillow and Wedge | Peanut Labor Ball
Number analyzed (Participants) | 69 | 70
minutes | 322.7 (174) | 331.3 (187.1)

3. Other Pre Specified Outcome: Third and Fourth Degree Lacerations
Description: Measuring if use of the Peanut Labor Ball impacts third and fourth degree lacerations during delivery
Time Frame: within the last 15-30 minutes of birth
Population: participants with vaginal delivery only
Measure: Count of Participants; unit: Participants
Arm/Group | Pillow and Wedge | Peanut Labor Ball
Number analyzed (Participants) | 69 | 70
Participants | 5 | 2

ADVERSE EVENTS:
Arm/Group | Pillow and Wedge | Peanut Labor Ball
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/91
Other Adverse Events (participants affected / at risk) | 0/100 | 0/91

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes